CLINICAL TRIAL: NCT06903299
Title: Utilisation of Tranexamic Acid in Elective Hip Arthroplasty
Brief Title: Prospective Investigation of Intra-Articular Tranexamic Acid Use in Elective Hip Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: 83V/2022 - AM
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-01

CONDITIONS: Blood Loss; Hemoglobin Change; Blood Transfusion; Heterotopic Ossification
MeSH Terms: conditions — Hemorrhage; Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Intra-articular Tranexamic acid application — Intra-articular Tranexamic acid application during THA and evaluation of postoperative blood losses, hemoglobin decline and associated blood transfusion, heterotopic ossification and other parameters.

SUMMARY:
Tranexamic acid (trans-4-aminomethyl cyclohexane carboxylic acid) is an antifibrinolytic substance that chemically belongs to the group of e-carboxylic acids. TXA is a synthetic amino acid derivative of lysine that competitively inhibits the activation of plasminogen to the serine protease, plasmin. TXA is a competitive inhibitor of tissue plasminogen activator, blocking the lysine-binding sites of plasminogen, resulting in inhibition of plasminogen activation and fibrin binding to plasminogen and therefore impairment of fibrinolysis.

Due to its antifibrinolytic effect (reduction of bleeding), TXA has been recently an increasing interest in orthopaedics, especially in elective major joint replacements.

The total hip arthroplasties (ΤΗΑ) are associated with perioperative blood losses exceeding 500 mL. Blood loss volumes are dependent on the chosen surgical approach and technique. Some patients that undergo elective hip replacement receive at least one blood unit in postoperative care. Heterotopic ossification is also a common complication after THA, presented as bone in soft tissue where bone normally does not appear. TXA reduces postoperative blood losses and consequently leads to less frequent blood transfusions. This has an impact on the economic burden for the health care system. Increased blood loss could lead to longer length of stay at the hospital and the connected economic consequences. TXA further reduces the incidence of heterotopic ossification after elective THA.

Objectives:

The aim of this study is to prospectively evaluate postoperative blood losses, hemoglobin decline and associated blood transfusion, heterotopic ossification and other parameters in patients with intraarticular application of Tranexamic acid during THA.

ELIGIBILITY:
Inclusion Criteria:

* Elective hip replacement

Exclusion Criteria:

* Traumatic hip replacement indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective hip replacement in the First Department of Orthopaedic Surgery, St. Anne's University Hospital, Brno, Czechia from 2023 to 2026.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Blood Loss | 48 hours postoperatively
  Total measured blood loss (in mL) within the first 24 to 48 hours after total hip arthroplasty (THA), calculated from surgical drains and hemoglobin change.

SECONDARY OUTCOMES:
Hemoglobin Change | Baseline, 24 hours, and 48 hours postoperatively
  Change in hemoglobin levels (g/dL) from preoperative baseline to 24 and 48 hours postoperatively. Change from baseline.
Incidence of Heterotopic Ossification | 1 year postoperatively
  Number of patients developing heterotopic ossification, assessed using radiographs at 6 weeks and 3 months postoperatively.
Incidence of Postoperative Complications | Up to 30 days postoperatively
  Number of patients experiencing complications such as deep vein thrombosis (DVT), pulmonary embolism (PE), wound infections, and other adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Orthopaedic Surgery, St. Anne's University Hospital and Faculty of Medicine, Masaryk University, Brno, Czechia, Brno, Czechia, Czechia